CLINICAL TRIAL: NCT01693770
Title: Primary Pain Palliation and Local Tumor Control in Bone Metastases Treated With Magnetic Resonance-guided Focused Ultrasound
Brief Title: Primary Pain Palliation in Bone Metastases Treated With Magnetic Resonance-guided Focused Ultrasound
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Alessandro Napoli, MD, PhD, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BM-MRgFUS
Record Dates: First submitted 2012-09-20; First posted 2012-09-26 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Secondary Malignant Neoplasm of Bone
Keywords: Bone Metastasis; Pain Palliation; High Intensity Focused Ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRgFUS (Other): High intensity focused ultrasound energy, delivered under the guidance of the MR images (MgFUS) allows for a predefined amount of energy to be delivered in the desired target (Metastasis). Bone readily absorbs focused ultrasound energy resulting in a thermo-related neurolysis of the periostium with consequent pain palliation. The amount of energy delivered can be modulated with the objective to penetrate cortical space and obtain necrosis of the metastasis thus preventing local recurrence.
  Interventions: Procedure: MRgFUS

INTERVENTIONS:
Procedure: MRgFUS — Focused ultrasound energy is accumulated into the target tissue (skeletal metastasis) thanks to the real time guidance of the MR images.
  Other Names: MRgFUS, ExAblate, InSightec; MR-HIFU; Magnetic Resonance-guided Focused Ultrasound

SUMMARY:
Magnetic Resonance guided Focused Ultrasound (MRgFUS) has demonstrated to be effective for pain control through thermally-induced cell death and periosteal denervation caused by cortical heating relative to acoustic energy absorption. There is also evidence that a high intensity focused ultrasound beam can penetrate through the cortical bone to the medullary space, producing thermal necrosis of cancer tissue. However, little is known about the potential effects of MRgFUS as first line therapeutic modality for pain palliation in skeletal metastases.

Our hypothesis sought to assess the clinical performance of MRgFUS primary treatment of painful bone metastases and determine the potential of this technique for local tumor control.

DETAILED DESCRIPTION:
Unlike previous studies, in which patients were enrolled for MRgFUS treatment because of the failure of other therapies, our study will be conducted in patients not previously treated with EBRT to the targeted lesion.

This is an important new feature, especially given the advantages of MRgFUS, such as lack of ionizing radiation, the ability to conduct treatment on an outpatient basis and the possibility to repeat the treatment as necessary.

ELIGIBILITY:
Inclusion Criteria:

* the presence of a known primary cancer and bone metastases confirmed by two or more imaging modalities;
* exhaustion or refusal of all other pain palliation methods including EBRT;
* confirmation of MRgFUS treatment feasibility at a preliminary MR planning examination (presence of an adequate acoustic window between the transducer, skin and target lesion and absence of bowel loops across the planned ultrasound path)

Exclusion Criteria:

* general contraindication to MR imaging (including pacemaker, ferromagnetic devices or implants)
* general contraindication to gadolinium-based contrast agents (intolerance and/or clinically proven chronic renal failure)
* general contraindication to general/epidural anesthesia or deep sedation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and efficacy of Magnetic Resonance-guided Focused Ultrasound (MRgFUS) for the primary treatment of painful bone metastases | 6 months
  Patients will be monitored for major or minor adverse events

SECONDARY OUTCOMES:
To correlate the treatment response to extent of tumor necrosis as determined by follow-up imaging | 6 months
  necrosis of the actual lesion will be analyzed according to area on non-perfused volume at the end of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Napoli, MD, PhD, Principal Investigator — Department of Radiological Sciences, Sapienza University of Rome
Locations (1):
- Policlinico Umberto I, Rome, Rome, Italy